CLINICAL TRIAL: NCT01328054
Title: A Phase IV, Placebo-controlled Single Sequence Crossover Study to Evaluate the Effect of Repeat Oral Doses of Lapatinib on Cardiac Repolarization in Patients With Advanced Cancer
Brief Title: A Study in Cancer Patients to Evaluate the Effect of Lapatinib on the QTc Interval
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 114271
Record Dates: First submitted 2011-03-10; First posted 2011-04-04 (Estimated); Results first posted 2016-06-08 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-05

CONDITIONS: Cancer
Keywords: cancer; cardiac repolarization; Holter monitor; pharmacokinetics; GW572016; lapatinib; QTc interval; safety; ECG
MeSH Terms: conditions — Neoplasms | interventions — Lapatinib

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- lapatinib/placebo (Experimental): This is a crossover study where subjects will receive placebo that mimics lapatinib for 2 days and lapatinib for 2 days. Subjects will not know when they are receiving placebo vs. lapatinib.
  Interventions: Drug: lapatinib; Drug: placebo matching lapatinib

INTERVENTIONS:
Drug: lapatinib — lapatinib commercial tablet, 2000mg, will be given as three separate doses (8 tablets/dose) given 12 hours apart over a 2 day period
Drug: placebo matching lapatinib — placebo matching lapatinib will be given as three separate doses (8 tablets/dose) given 12 hours apart over a 2 day period

SUMMARY:
This study will estimate the effect of lapatinib on cardiac repolarization (QTc interval duration) in subjects with advanced solid tumors. The study treatment period will occur over five days and an End of Study visit will be conducted on Day 8 (or no later than 3 days beyond Day 8). Subjects will receive placebo that mimics lapatinib for 2 days as three separate doses given 12 hours apart (8 tablets/dose) and lapatinib (2000mg) for 2 days as three separate doses given 12 hours apart (8 tablets/dose). Subjects will not know when they are receiving placebo vs. lapatinib. Digital 12-lead ECG recordings will be extracted from continuous ECG recordings obtained via a Holter monitor to measure QTc interval duration. Triplicate ECG measurements of QTc interval will be taken at pre-specified times at Day 1 (Baseline) and pre-dose and up to 24 hours after the third dose of placebo or lapatinib on Study Days 2 and 4. Pharmacokinetic sampling will occur immediately following each pre-specified QTc measurement in subjects dosed with placebo or lapatinib. Subjects who complete participation in this study, if they are eligible, will be offered the option to continue treatment with lapatinib, either alone or in combination with other oncology drugs in pre-selected anticancer regimens, in a continuation protocol, EGF111767.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of: Metastatic breast cancer that over-expresses ErbB2 OR Recurrent, advanced, or metastatic solid tumor malignancy (including breast cancer that does not over-express ErbB2) that is refractory to standard therapies, for which there is no approved therapy, or for which lapatinib in combination with one of the permitted anti-cancer regimens specified in the continuation study EGF111767 may provide clinical benefit.
* A female subject must be of non-childbearing potential or willing to use acceptable contraception.
* A male subject with a female partner of childbearing potential must agree to use acceptable contraception.
* Is able to swallow and retain oral medication and does not have uncontrolled emesis.
* ECOG performance status 0 to 1.
* Adequate bone marrow function: ANC (absolute neutrophil count) >/=1.5 x 10^9/L, Hemoglobin >/=9 g/dL, Platelets >/=75 x 10^9/L.
* Albumin >/=3 g/dL.
* Serum bilirubin </=1.5 x ULN.
* AST and ALT </=3 x ULN .
* Serum Creatinine </=1.5 mg/dL or Calculated Creatinine Clearance >/= 50 mL/min.
* Serum potassium and magnesium levels within normal limits.
* Has a LVEF within the normal institutional range (or >/=50%).

Exclusion Criteria:

* Any of the following ECG findings: QTcF interval >480 msec, PR interval >240 msec or </=110 msec, Bradycardia defined as sinus rate <50 beats per minute.
* Cardiac conduction abnormalities denoted by any of the following: Evidence of second-degree (type II) or third-degree atrioventricular block, Evidence of ventricular pre-excitation, Electrocardiographic evidence of complete left bundle branch block (LBBB), Intraventricular conduction delay with QRS duration >120 msec, Atrial fibrillation, Presence of cardiac pacemaker.
* History of any one of the following cardiovascular conditions within the past 6 months: Class III or IV congestive heart failure as defined by the New York Heart Association (NYHA), cardiac angioplasty or stenting, myocardial infarction, unstable angina, symptomatic peripheral vascular disease or other clinically significant cardiac disease.
* Personal history of long-QT syndrome.
* Is pregnant or lactating.
* Has malabsorption syndrome, or has undergone a resection or bypass of the distal stomach and pylorus, or small bowel.
* Has acute or currently active/requiring anti-viral therapy hepatic or biliary disease (with the exception of subjects with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment).
* Has evidence of symptomatic or uncontrolled brain metastases or leptomeningeal disease. Subjects with brain metastases treated by surgery and/or radiotherapy are eligible if neurologically stable and do not require steroids or anticonvulsants for at least 28 days prior to the first dose of study drug.
* Has known immediate or delayed hypersensitivity reaction or idiosyncratic reaction to drugs chemically related to the investigational product.
* Has received anti-cancer therapy (including chemotherapy, radiation therapy, immunotherapy, biologic therapy, investigational therapy, surgery, or hormonal therapy) within 14 days prior to the first dose of study medication.
* Is receiving any prohibited medication or consuming any food or beverage within the timeframe indicated on the prohibited medication list in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2011-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- United States (4):
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Lebanon, New Hampshire
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Salt Lake City, Utah

REFERENCES:
- [Derived] Coker SA, Hurwitz HI, Sharma S, Wang D, Jordaan P, Zarate JP, Lewis LD. The effects of lapatinib on cardiac repolarization: results from a placebo controlled, single sequence, crossover study in patients with advanced solid tumors. Cancer Chemother Pharmacol. 2019 Aug;84(2):383-392. doi: 10.1007/s00280-019-03880-9. Epub 2019 Jun 11. PMID 31187169

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants (par.) underwent screening assessments within 14 days prior to the start of study treatment to determine their eligibility for enrollment. Study treatment was administered over a period of 5 days, and an End of Study visit was conducted on Day 8-11.
Groups:
- Placebo: Participants received three doses of matching placebo in the morning and evening on Day 1 and in the morning on Day 2.
- Lapatinib 2000 mg: Participants received three doses of lapatinib 2000 milligrams (mg) (250 mg x 8 tablets/dose) in the morning and evening on Day 3 and in the morning on Day 4.
Period: Placebo on Day 1 and Day 2 (2 Days)
Arm/Group | Placebo | Lapatinib 2000 mg
Started | 57 | 0
Completed | 57 | 0
Not Completed | 0 | 0
Period: Lapatinib on Day 3 and Day 4 (2 Days)
Arm/Group | Placebo | Lapatinib 2000 mg
Started | 0 | 58 (One par. was double dosed with lapatinib due to a dosing error - reason for difference in # Started.)
Completed | 0 | 53
Not Completed | 0 | 5
Not completed — Adverse Event | 0 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Placebo and Lapatinib 2000 mg: Participants received three doses of matching placebo in the morning and evening on Day 1 and in the morning on Day 2. Participants then received three doses of lapatinib 2000 mg (250 mg x 8 tablets/dose) in the morning and evening on Day 3 and in the morning on Day 4.
Arm/Group | Placebo and Lapatinib 2000 mg
Number analyzed (Participants) | 58
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.1 (12.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 21
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 3
  Asian - East Asian Heritage | 1
  Asian - South East Asian Heritage | 1
  White - White/Caucasian/European Heritage | 51
  missing | 2

OUTCOME MEASURES:

1. Primary Outcome: Treatment Difference in Duration of Cardiac Ventricular Depolarization and Repolarization Interval (QT) in Fridericia-corrected QT Interval (QTcF) Values Between Placebo and Lapatinib 2000mg
Description: A Holter monitor is an ambulatory portable device used for continuously monitoring the cardiovascular system. Three replicate electrocardiograms (ECGs) were collected at 30, 15, and 0 minutes prior to the administration of study treatment (trt) on Days 1 and 3 and pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, and 24 hr post-dose on Days 2 and 4. The 3 readings at each time point (TP) were averaged prior to any analysis. BL is the average of the pre-dose QTcF values (triplicate) taken on Day 1 for PBO and on Day 3 for LAP. Mean change from BL was calculated by subtracting the BL values from individual QTcF for each TP. BL adjusted mean difference in absolute QTcF between LAB and PBO (trt difference) with the corresponding 90% confidence interval (CI) was estimated for each TP (pre-dose and 1, 2, 3, 4, 6, 8, 10, 12, and 24-hr post-dose). Trt difference analysis was performed by a repeated measures analysis of variance adjusted for trt group, TP, and trt group*TP interaction.
Time Frame: Baseline (BL) (Day1) and pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, and 24-hours (hr) post-dose on Day 2 for placebo (PBO). Baseline (Day 3) and pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, and 24-hours post-dose on Day 4 for lapatinib (LAP).
Population: Evaluable Population: all participants in the All-Treated Subjects (ATS) Population who met the criteria for dosing compliance, ECG acquisition, and Baseline ECG acquisition. The ATS Population is comprised of all participants who received at least one dose of study medication (placebo or lapatinib).
Measure: Least Squares Mean (Standard Error); unit: Milliseconds
Groups:
- Lapatinib 2000 mg: Participants received three doses of lapatinib 2000 mg (250 mg x 8 tablets/dose) in the morning and evening on Day 3 and in the morning on Day 4.
Arm/Group | Placebo | Lapatinib 2000 mg
Number analyzed (Participants) | 37 | 37
Milliseconds
  Pre-dose | -3.71 (1.53) | 2.60 (1.53)
  1 hour | 0.66 (1.46) | 7.09 (1.47)
  2 hour | 0.49 (1.23) | 8.20 (1.24)
  3 hour | 2.78 (1.48) | 9.19 (1.48)
  4 hour | 3.18 (1.73) | 9.78 (1.73)
  6 hour | -4.50 (1.82) | 1.36 (1.83)
  8 hour | -5.09 (1.93) | -0.18 (1.95)
  10 hour | -4.53 (1.98) | 4.22 (1.99)
  12 hour | -1.49 (1.96) | 4.27 (1.96)
  24 hour | -1.25 (1.52) | 2.51 (1.55)
Statistical Analysis 1: Comparison: Placebo vs Lapatinib 2000 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 6.31, 90% CI 2-sided [2.72 to 9.89], Standard Error of Mean 2.151 — Confidence interval (CI), estimated value and dispersion value of is presented for pre dose
Statistical Analysis 2: Comparison: Placebo vs Lapatinib 2000 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 6.43, 90% CI 2-sided [3.00 to 9.87], Standard Error of Mean 2.059 — CI, estimated value and dispersion value of is presented for 1 hour post dose
Statistical Analysis 3: Comparison: Placebo vs Lapatinib 2000 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 7.71, 90% CI 2-sided [4.82 to 10.60], Standard Error of Mean 1.734 — CI, estimated value and dispersion value of is presented for 2 hour post dose
Statistical Analysis 4: Comparison: Placebo vs Lapatinib 2000 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 6.42, 90% CI 2-sided [2.94 to 9.89], Standard Error of Mean 2.085 — CI, estimated value and dispersion value of is presented for 3 hour post dose
Statistical Analysis 5: Comparison: Placebo vs Lapatinib 2000 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 6.60, 90% CI 2-sided [2.54 to 10.65], Standard Error of Mean 2.434 — CI, estimated value and dispersion value of is presented for 4 hour post dose
Statistical Analysis 6: Comparison: Placebo vs Lapatinib 2000 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 5.86, 90% CI 2-sided [1.57 to 10.14], Standard Error of Mean 2.573 — CI, estimated value and dispersion value of is presented for 6 hour post dose
Statistical Analysis 7: Comparison: Placebo vs Lapatinib 2000 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 4.91, 90% CI 2-sided [0.35 to 9.47], Standard Error of Mean 2.735 — CI, estimated value and dispersion value of is presented for 8 hour post dose
Statistical Analysis 8: Comparison: Placebo vs Lapatinib 2000 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 8.75, 90% CI 2-sided [4.08 to 13.42], Standard Error of Mean 2.800 — CI, estimated value and dispersion value of is presented for 10 hour post dose
Statistical Analysis 9: Comparison: Placebo vs Lapatinib 2000 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 5.76, 90% CI 2-sided [1.16 to 10.36], Standard Error of Mean 2.759 — CI, estimated value and dispersion value of is presented for 12 hour post dose
Statistical Analysis 10: Comparison: Placebo vs Lapatinib 2000 mg; Test type: Superiority or Other; Mean Difference (Final Values) = 3.75, 90% CI 2-sided [0.15 to 7.36], Standard Error of Mean 2.164 — CI, estimated value and dispersion value of is presented for 24 hour post dose

2. Secondary Outcome: Change From Baseline in the Holter ECG Parameters of QT Interval, Corrected QT Interval (QTc), Bazett Corrected QTc Interval (QTcB), Individual-corrected QT Interval (QTcI), RR Interval, PR Interval, and QRS Duration at Indicated Time Points
Description: A Holter monitor is an ambulatory portable device for continuously monitoring the cardiovascular system. Change from Baseline in QT interval, QTc interval, QTcB interval, QTcI interval, RR interval, PR interval, and QRS duration at each time point for lapatinib was assessed in comparison with time-matched placebo. Three replicate ECGs were collected at 30, 15, and 0 minutes prior to the administration of study treatment on Days 1 and 3 and pre-dose and 1, 2, 3, 4, 6, 8, 10, and 24 hours post dose on Days 2 and 4. The three readings at each time point were averaged prior to any analysis. Baseline is the average of the pre-dose ECGs (triplicate) taken on Day 1 for placebo and Day 3 for lapatinib. Change from Baseline was calculated by subtracting the Baseline values from individual post-Baseline values for each time point.
Time Frame: Baseline (Day1) and pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, and 24-hours post-dose on Day 2 for placebo. Baseline (Day 3) and pre-dose, 1, 2, 3, 4, 6, 8, 10, 12, and 24-hours post-dose on Day 4 for lapatinib.
Population: Evaluable Population. Only participants available at the specified time point (represented as n=X, X in the category title) were analyzed.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Placebo | Lapatinib 2000 mg
Number analyzed (Participants) | 37 | 37
Milliseconds
  QT interval (predose), n=37, 37 | -6.24 (16.788) | 1.05 (17.033)
  QT interval (1 hour), n=37, 37 | 0.10 (15.320) | 7.69 (18.870)
  QT interval (2 hour), n=37, 37 | 1.24 (15.055) | 10.66 (16.315)
  QT interval (3 hour), n=37, 37 | 2.14 (14.798) | 11.09 (18.805)
  QT interval (4 hour), n=37, 37 | 1.14 (16.741) | 10.09 (20.062)
  QT interval (6 hour), n=37, 36 | -17.77 (21.240) | -6.97 (20.888)
  QT interval (8 hour), n=37, 36 | -13.51 (20.997) | -6.88 (25.718)
  QT interval (10 hour), n=37, 37 | -15.99 (19.617) | -3.68 (21.191)
  QT interval (12 hour), n=37, 37 | -11.28 (18.576) | -1.58 (21.615)
  QT interval (24 hour), n=37, 35 | -4.10 (15.152) | 0.54 (17.928)
  QTcI interval (predose), n=37, 37 | -6.40 (13.133) | 2.24 (12.930)
  QTcI interval (1 hour), n=37, 37 | -1.45 (10.925) | 6.00 (13.053)
  QTcI interval (2 hour), n=37, 37 | -1.40 (12.037) | 8.42 (13.054)
  QTcI interval (3 hour), n=37, 37 | -0.05 (12.015) | 8.76 (14.227)
  QTcI interval (4 hour), n=37, 37 | 0.32 (13.786) | 8.00 (15.274)
  QTcI interval (6 hour), n=37, 36 | -11.53 (15.688) | -3.86 (14.987)
  QTcI interval (8 hour), n=37, 36 | -10.13 (14.223) | -4.65 (17.336)
  QTcI interval (10 hour), n=37, 37 | -11.70 (16.374) | -0.26 (16.461)
  QTcI interval (12 hour), n=37, 37 | -6.22 (17.752) | 0.35 (15.458)
  QTcI interval (24 hour), n=37, 35 | -4.71 (9.677) | 2.03 (13.715)
  QTcB interval (predose), n=37, 37 | -2.18 (10.942) | 4.07 (9.271)
  QTc B interval (1 hour), n=37, 37 | 1.07 (8.061) | 7.37 (8.978)
  QTcB interval (2 hour), n=37, 37 | 0.11 (8.918) | 7.43 (8.626)
  QTcB interval (3 hour), n=37, 37 | 3.13 (8.954) | 8.77 (8.846)
  QTcB interval (4 hour), n=37, 37 | 4.38 (10.786) | 10.14 (9.334)
  QTcB interval (6 hour), n=37, 36 | 3.11 (10.275) | 7.08 (12.382)
  QTcB interval (8 hour), n=37, 36 | -0.29 (11.117) | 3.97 (10.481)
  QTcB interval (10 hour), n=37, 37 | 1.93 (9.871) | 9.25 (13.060)
  QTcB interval (12 hour), n=37, 37 | 4.21 (10.238) | 8.08 (11.379)
  QTcB interval (24 hour), n=37, 35 | 0.42 (8.756) | 5.38 (7.752)
  RR interval (predose), n=37, 37 | -19.19 (78.141) | -9.68 (74.332)
  RR interval (1 hour), n=37, 37 | -5.38 (65.333) | 3.14 (78.012)
  RR interval (2 hour), n=37, 37 | 2.71 (72.996) | 16.07 (63.665)
  RR interval (3 hour), n=37, 37 | -5.38 (67.323) | 12.50 (67.526)
  RR interval (4 hour), n=37, 37 | -13.43 (64.043) | 2.90 (78.299)
  RR interval (6 hour), n=37, 36 | -85.20 (93.003) | -61.77 (83.279)
  RR interval (8 hour), n=37, 36 | -54.95 (92.426) | -41.60 (90.545)
  RR interval (10 hour), n=37, 37 | -74.17 (82.639) | -49.38 (75.999)
  RR interval (12 hour), n=37, 37 | -63.20 (79.552) | -38.38 (74.737)
  RR interval (24 hour), n=37, 35 | -19.69 (67.199) | -17.15 (69.927)
  PR interval (predose), n=37, 37 | -1.87 (9.162) | 3.48 (6.000)
  PR interval (1 hour), n=37, 37 | -0.20 (7.026) | 4.90 (8.492)
  PR interval (2 hour), n=37, 37 | 0.90 (6.563) | 4.98 (8.952)
  PR interval (3 hour), n=37, 37 | 0.25 (7.839) | 4.86 (7.668)
  PR interval (4 hour), n=37, 37 | -0.40 (7.321) | 4.05 (7.713)
  PR interval (6 hour), n=37, 36 | -3.05 (9.165) | 0.32 (8.815)
  PR interval (8 hour), n=37, 36 | -2.72 (6.993) | 0.10 (9.325)
  PR interval (10 hour), n=37, 37 | -4.77 (6.892) | -0.23 (8.743)
  PR interval (12 hour), n=37, 37 | -2.97 (7.071) | 1.81 (9.503)
  PR interval (24 hour), n=37, 35 | -1.61 (7.433) | 0.94 (6.388)
  QRS interval (predose), n=37, 37 | 0.88 (3.562) | 0.46 (3.860)
  QRS interval (1 hour), n=37, 37 | 1.45 (3.766) | 0.67 (4.164)
  QRS interval (2 hour), n=37, 37 | 1.08 (3.290) | 0.66 (3.851)
  QRS interval (3 hour), n=37, 37 | 0.89 (3.896) | 1.03 (4.786)
  QRS interval (4 hour), n=37, 37 | 1.17 (3.612) | 1.83 (4.617)
  QRS interval (6 hour), n=37, 36 | 0.88 (3.839) | 1.65 (4.212)
  QRS interval (8 hour), n=37, 36 | 0.80 (3.500) | 1.47 (5.417)
  QRS interval (10 hour), n=37, 37 | 0.70 (3.574) | 1.48 (5.042)
  QRS interval (12 hour), n=37, 37 | 0.13 (3.634) | 1.92 (3.992)
  QRS interval (24 hour), n=37, 35 | 1.07 (3.890) | 0.97 (3.461)

3. Secondary Outcome: Number of Participants With 12-lead Holter ECG Findings at the Indicated Time Points
Description: The number of participants with 12-lead Holter ECG findings of normal (NL), abnormal not clinically significant (Abn NCS), and abnormal clinically significant (Abn CS) are reported. Abnormal ECG findings or change in ECG morphological patterns were based on the ECG interpretations provided by the ECG core lab. Three replicate 12-lead Holter ECGs were collected at -30, -15, and 0 minutes prior to the administration of study treatment on Days 1 (Baseline for placebo) and 3 (Baseline for lapatinib) and pre-dose and 1, 2, 3, 4, 6, 8, 10,12, and 24 hours post dose on Days 2 and 4. The three readings at each time point were averaged prior to any analysis. Baseline is the pre-dose ECGs (triplicate) taken on Day 1 for placebo and on Day 3 for lapatinib.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Placebo | Lapatinib 2000 mg
Number analyzed (Participants) | 37 | 37
Participants
  -30 minutes (NL), n=35, 32 | 35 | 32
  -30 minutes (Abn NCS), n=35, 32 | 0 | 0
  -30 minutes (Abn CS), n=35, 32 | 0 | 0
  -15 minutes (NL), n=34, 32 | 34 | 32
  -15 minutes (Abn NCS), n=34, 32 | 0 | 0
  -15 minutes (Abn CS), n=34, 32 | 0 | 0
  0 minutes (NL), n=34, 32 | 34 | 32
  0 minutes (Abn NCS), n=34, 32 | 0 | 0
  0 minutes (Abn CS), n=34, 32 | 0 | 0
  Pre dose (NL), n=33, 31 | 33 | 31
  Pre dose (Abn NCS), n=33, 31 | 0 | 0
  Pre dose (Abn CS), n=33, 31 | 0 | 0
  1 hour (NL), n=33, 30 | 33 | 30
  1 hour (Abn NCS), n=33, 30 | 0 | 0
  1 hour (Abn CS), n=33, 30 | 0 | 0
  2 hour (NL), n=31, 28 | 31 | 28
  2 hour (Abn NCS), n=31, 28 | 0 | 0
  2 hour (Abn CS), n=31, 28 | 0 | 0
  3 hour (NL), n=31, 27 | 31 | 27
  3 hour (Abn NCS), n=31, 27 | 0 | 0
  3 hour (Abn CS), n=31, 27 | 0 | 0
  4 hour (NL), n=34, 28 | 34 | 28
  4 hour (Abn NCS), n=34, 28 | 0 | 0
  4 hour (Abn CS), n=34, 28 | 0 | 0
  6 hour (NL), n=31, 27 | 31 | 27
  6 hour (Abn NCS), n=31, 27 | 0 | 0
  6 hour (Abn CS), n=31, 27 | 0 | 0
  8 hour (NL), n=31, 27 | 31 | 27
  8 hour (Abn NCS), n=31, 27 | 0 | 0
  8 hour (Abn CS), n=31, 27 | 0 | 0
  10 hour (NL), n=32, 31 | 32 | 31
  10 hour (Abn NCS), n=32, 31 | 0 | 0
  10 hour (Abn CS), n=32, 31 | 0 | 0
  12 hour (NL), n=31, 29 | 31 | 29
  12 hour (Abn NCS), n=31, 29 | 0 | 0
  12 hour (Abn CS), n=31, 29 | 0 | 0
  24 hour (NL), n=0, 27 | 0 | 27
  24 hour (Abn NCS), n=0, 27 | 0 | 0
  24 hour (Abn CS), n=0, 27 | 0 | 0

4. Secondary Outcome: Number of Participants With the Worst-case Post-Baseline 12-lead Holter ECG Findings With Significant ST, T Wave, and U Wave Abnormalities
Description: Abnormal ECG findings or change in ECG morphological patterns were based on the ECG interpretations provided by the ECG core lab. Three replicate Holter ECGs were collected at 30, 15, and 0 minutes prior to the administration of study treatment on Days 1 (Baseline for placebo) and 3 (Baseline for lapatinib) and pre-dose and 1, 2, 3, 4, 6, 8, 10, and 24 hours post dose on Days 2 and 4. The three readings at each time point were averaged prior to any analysis. Baseline is the pre-dose ECGs (triplicate) taken on Day 1 for placebo and Day 3 for lapatinib. The number of participants with the worst-case post-Baseline 12-lead Holter ECG findings with significant ST, T wave, and U wave abnormalities were analyzed.
Time Frame: as for outcome 2
Population: Pharmacodynamic (PD) Population: all participants from the All Treated Subjects Population (ATS) who completed the ECG acquisition via Holter monitoring of at least one time point on Days 1, 2, 3 and 4.
Measure: Number; unit: Participants
Arm/Group | Placebo | Lapatinib 2000 mg
Number analyzed (Participants) | 51 | 52
Participants | 11 | 14

5. Secondary Outcome: Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE)
Description: An AE is defined as any untoward medical occurrence in a participant temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity or is a congenital anomaly/birth defect, or is an important medical eventsthat jeopardizes the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in the above definition, new primary cancers, liver events, cardiac dysfunction, pneumonitis, and laboratory abnormalities.
Time Frame: From the start of study treatment until follow-up (within approximately 28 days following the last dose of study medication [up to end of Study Week 4])
Population: ATS Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Lapatinib 2000 mg
Number analyzed (Participants) | 57 | 58
Participants
  Any AE | 16 | 44
  Any SAEs | 0 | 4

6. Secondary Outcome: Mean Albumin, and Hemoglobin at the Indicated Time Points
Description: Blood samples were collected for the measurement of albumin and hemoglobin at Baseline; Days 5 and 8-11. Baseline is defined as the most recent, non-missing value from a central laboratory prior to or on the first study treatment dose date.
Time Frame: Baseline; Day 5 and end of study visit on Day 8-11
Population: ATS Population. Only participants available at the specified time point (represented as n=X in the category title) were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Groups:
- Placebo/Lapatinib 2000 mg: Participants received three doses of matching placebo in the morning and evening on Day 1 and in the morning on Day 2. Participants then received three doses of lapatinib 2000 mg (250 mg x 8 tablets/dose) in the morning and evening on Day 3 and in the morning on Day 4.
Arm/Group | Placebo/Lapatinib 2000 mg
Number analyzed (Participants) | 58
Grams per liter (g/L)
  Albumin (Baseline), n=58 | 38.8 (3.83)
  Albumin (Day 5), n=49 | 35.5 (4.42)
  Albumin (Day 8-11), n=55 | 37.5 (3.94)
  Hemoglobin (Baseline), n=58 | 123.7 (15.45)
  Hemoglobin (Day 5), n=48 | 114.8 (15.63)
  Hemoglobin (Day 8-11), n=55 | 117.6 (15.51)

7. Secondary Outcome: Mean Alkaline Phosphatase (ALP), Alanine Aminotransferase (ALT), and Aspartate Aminotransferase (AST) at the Indicated Time Points
Description: Blood samples were collected for the measurement of ALP, ALT, and AST at Baseline; Days 5 and 8-11. Baseline is defined as the most recent, non-missing value from a central laboratory prior to or on the first study treatment dose date.
Time Frame: Baseline; Day 5 and end of study visit on Day 8-11
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Groups:
- Placebo/Lapatinib 2000mg: Participants received three doses of matching placebo in the morning and evening on Day 1 and in the morning on Day 2. Participants then received three doses of lapatinib 2000 mg (250 mg x 8 tablets/dose) in the morning and evening on Day 3 and in the morning on Day 4.
Arm/Group | Placebo/Lapatinib 2000mg
Number analyzed (Participants) | 58
International units per liter (IU/L)
  ALP (baseline), n=58 | 116.9 (90.91)
  ALP (Day 5), n=49 | 111.2 (97.55)
  ALP (Day 8-11), n=55 | 116.7 (107.50)
  ALT (baseline), n=58 | 25.9 (17.09)
  ALT (Day 5), n=49 | 23.1 (14.85)
  ALT (Day 8-11), n=55 | 24.2 (16.98)
  AST (baseline), n=58 | 29.7 (16.09)
  AST (Day 5), n=48 | 26.9 (14.16)
  AST (Day 8-11), n=55 | 30.3 (16.46)

8. Secondary Outcome: Mean Direct Bilirubin, Total Bilirubin, and Creatinine at the Indicated Time Points
Description: Blood samples were collected for the measurement of direct bilirubin, total bilirubin, and creatinine at Baseline; Days 5 and 8-11; Baseline is defined as the most recent, non-missing value from a central laboratory prior to or on the first study treatment dose date.
Time Frame: Baseline; Day 5 and end of study visit on Day 8-11
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Micromoles per liter (µmol/L)
Arm/Group | Placebo/Lapatinib 2000mg
Number analyzed (Participants) | 58
Micromoles per liter (µmol/L)
  Direct Bilirubin (Baseline), n=58 | 2.683 (1.6678)
  Direct Bilirubin (Day 5), n=46 | 3.123 (2.0490)
  Direct Bilirubin (Day 8-11), n=54 | 2.502 (1.4749)
  Bilirubin (Baseline), n=58 | 10.496 (4.3620)
  Bilirubin (Day 5), n=49 | 13.450 (6.2571)
  Bilirubin (Day 8-11), n=55 | 9.980 (4.8786)
  Creatinine (Baseline), n=58 | 73.448 (23.6266)
  Creatinine (Day 5), n=49 | 77.124 (27.9006)
  Creatinine (Day 8-11), n=55 | 74.192 (25.0945)

9. Secondary Outcome: Mean Calcium, Chloride, Carbon Dioxide (CO2), Potassium, Sodium, Magnesium and Urea at the Indicated Time Points
Description: Blood samples were collected for the measurement of calcium, chloride, CO2, potassium, sodium, magnesium and urea at Baseline; at Days 5 and 8-11. Baseline is defined as the most recent, non-missing value from a central laboratory prior to or on the first study treatment dose date.
Time Frame: Baseline; Day 5 and end of study visit on Day 8-11
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Placebo/Lapatinib 2000 mg
Number analyzed (Participants) | 58
Millimoles per liter (mmol/L)
  Calcium (Baseline), n=57 | 2.344 (0.1176)
  Calcium (Day 5), n=49 | 2.231 (0.1148)
  Calcium (Day 8-11), n=55 | 2.303 (0.1336)
  Chloride (Baseline), n=58 | 103.6 (3.42)
  Chloride (Day 5), n=49 | 104.4 (2.76)
  Chloride (Day 8-11), n=55 | 104.7 (3.03)
  CO2 (Baseline), n=57 | 26.965 (2.7449)
  CO2 (Day 5), n=49 | 26.053 (3.1032)
  CO2 (Day 8-11), n=55 | 26.345 (2.9390)
  Potassium (Baseline), n=58 | 4.05 (0.337)
  Potassium (Day 5), n=49 | 3.84 (0.425)
  Potassium (Day 8-11), n=55 | 3.98 (0.372)
  Sodium (Baseline), n=58 | 138.8 (2.42)
  Sodium (Day 5), n=49 | 138.5 (2.34)
  Sodium (Day 8-11), n=55 | 139.0 (2.55)
  Magnesium (Baseline), n=58 | 0.835 (0.0906)
  Magnesium (Day 5, n=49) | 0.769 (0.1420)
  Magnesium (Day 8-11), n=55 | 0.795 (0.1088)
  Urea (Baseline), n=58 | 5.273 (1.9485)
  Urea (Day 5), n=49 | 5.078 (1.7032)
  Urea (Day 8-11), n=55 | 5.095 (1.7922)

10. Secondary Outcome: Mean Total Neutrophils (ANC [Absolute Neutrophil Count]), Platelets and Leukocyte Count at the Indicated Time Points
Description: Blood samples were collected for the measurement of total neutrophils (ANC), platelets, and leukocyte count at Baseline; Days 5 and 8-11. Baseline was defined as the most recent, non-missing value from a central laboratory prior to or on the first study treatment dose date.
Time Frame: Baseline; Day 5 and end of study visit on Day 8-11
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter (GI/L)
Groups:
- Placebo/ Lapatinib: Participants received three doses of matching placebo in the morning and evening on Day 1 and in the morning on Day 2. Participants then received three doses of lapatinib 2000 mg (250 mg x 8 tablets/dose) in the morning and evening on Day 3 and in the morning on Day 4.
Arm/Group | Placebo/ Lapatinib
Number analyzed (Participants) | 58
10^9 cells per liter (GI/L)
  ANC (Baseline), n=58 | 23.959 (30.0190)
  ANC (Day 5), n=48 | 25.802 (30.8866)
  ANC (Day 8-11), n=55 | 23.848 (29.8574)
  Platelets (Baseline), n=58 | 262.6 (90.29)
  Platelets (Day 5), n=48 | 239.3 (86.90)
  Platelets (Day 8-11), n=55 | 263.7 (92.44)
  Leukocytes (Baseline), n=58 | 6.686 (2.5192)
  Leukocytes (Day 5), n=48 | 6.227 (2.3865)
  Leukocytes (Day 8-11), n=55 | 7.198 (3.6319)

11. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at the Indicated Time Points
Description: Blood pressure measurements included SBP and DBP and were obtained at Baseline; on Day 2 (at pre-dose, 4, 8, 12 and 24 hours post dose), and on Day 4 (at pre-dose, 4, 8, 12 and 24 hours post dose). Baseline is defined as the most recent, non-missing value prior to or on the first study treatment dose date. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; on Day 2 (at pre-dose, 4, 8, 12 and 24 hours post-dose), and on Day 4 (at pre-dose, 4, 8, 12 and 24 hours post-dose)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Millimeter of mercury (mmHg)
Arm/Group | Placebo/Lapatinib 2000 mg
Number analyzed (Participants) | 58
Millimeter of mercury (mmHg)
  Systolic BP (Day 2-Pre dose), n=58 | -3.5 (13.19)
  Systolic BP (Day 2-4 hour post dose), n=58 | -2.1 (13.21)
  Systolic BP (Day 2-8 hour post dose), n=58 | -7.0 (13.71)
  Systolic BP (Day 2-12 hour post dose), n=58 | -4.2 (14.62)
  Systolic BP (Day 2-24 hour post dose), n=58 | -2.2 (11.29)
  Systolic BP (Day 4-Pre dose), n=56 | -9.4 (14.55)
  Systolic BP (Day 4-4 hour post dose), n=55 | -8.7 (12.75)
  Systolic BP (Day 4-8 hour post dose), n=55 | -8.3 (14.15)
  Systolic BP (Day 4-12 hour post dose), n=54 | -8.8 (13.26)
  Systolic BP (Day 4-24 hour post dose), n=54 | -4.8 (11.54)
  Diastolic BP (Day 2-Pre dose), n=58 | -4.2 (8.34)
  Diastolic BP (Day 2-4 hour post dose), n=58 | -4.6 (8.13)
  Diastolic BP (Day 2-8 hour post dose), n=58 | -8.2 (9.13)
  Diastolic BP (Day 2-12 hour post dose), n=58 | -6.3 (8.77)
  Diastolic BP (Day 2-24 hour post dose), n=58 | -2.9 (7.27)
  Diastolic BP (Day 4-Pre dose), n=56 | -8.6 (8.06)
  Diastolic BP (Day 4-4 hour post dose), n=55 | -7.3 (8.49)
  Diastolic BP (Day 4-8 hour post dose), n=55 | -7.4 (10.12)
  Diastolic BP (Day 4-12 hour post dose), n=54 | -8.1 (9.29)
  Diastolic BP (Day 4-24 hour post dose), n=54 | -5.0 (8.14)

12. Secondary Outcome: Change From Baseline in Heart Rate at the Indicated Time Points
Description: Heart rate were measured at Baseline; on Day 2 (at pre-dose, 4, 8, 12 and 24 hours post dose), and on Day 4 (at pre-dose, 4, 8, 12 and 24 hours post dose. Baseline is defined as the most recent, non-missing value prior to or on the first study treatment dose date. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; on Day 2 (at pre-dose, 4, 8, 12 and 24 hours post dose), and on Day 4 (at pre-dose, 4, 8, 12 and 24 hours post dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo/Lapatinib 2000 mg
Number analyzed (Participants) | 58
Beats per minute
  Day 2-Pre dose, n=57 | 3.9 (9.82)
  Day 2-4 hour post dose, n=58 | -1.7 (9.10)
  Day 2-8 hour post dose, n=58 | 3.2 (9.96)
  Day 2-12 hour post dose, n=58 | 3.3 (10.02)
  Day 2-24 hour post dose, n=58 | 0.8 (9.78)
  Day 4-Pre dose, n=56 | 3.5 (10.88)
  Day 4-4 hour post dose, n=55 | -2.0 (10.89)
  Day 4-8 hour post dose, n=55 | 2.5 (11.12)
  Day 4-12 hour post dose, n=54 | 3.2 (11.09)
  Day 4-24 hour post dose, n=54 | 1.8 (8.75)

13. Secondary Outcome: Number of Participants With 12-lead ECG Findings at Indicated Time Points
Description: The number of participants with the 12-lead ECG findings normal (NL), abnormal not clinically significant (Abn NCS), and abnormal clinically significant (Abn CS) are reported. Clinical significance was based on the medical and scientific judgement of the investigator or qualified designee. A single safety 12-lead ECG was performed using a standard 12-lead ECG machine at Baseline; on Day 1 (at pre-dose); on Day 2 (at pre-dose, 4, 8, 12 and 24 hours post-last- dose); on Day 4 (at pre-dose, 4, 8, 12 and 24 hours post-last-dose); at the End of Study visit (Day 8-11); and at the post-treatment Follow-up visit (if applicable).
Time Frame: BL;Day 1 (at pre-dose);Day 2 (at pre-dose, 4, 8, 12 and 24 hr post dose);Day 4 (at pre-dose, 4, 8, 12 and 24 hr post dose);End of Study visit (Day 8-11); and Follow-up (within approx 28 days following last dose of study trt [up to end of Study Week 4])
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Placebo/Lapatinib 2000 mg
Number analyzed (Participants) | 58
Participants
  Baseline (NL), n=58 | 36
  Baseline (Abn NCS), n=58 | 22
  Baseline (Abn CS), n=58 | 0
  Day 1 (NL), n=58 | 35
  Day 1 (Abn NCS), n=58 | 23
  Day 1 (Abn CS), n=58 | 0
  Day 2 (Pre dose) (NL), n=58 | 32
  Day 2 (Pre dose) (Abn NCS), n=58 | 26
  Day 2 (Pre dose) (Abn CS), n=58 | 0
  Day 2 (4 hours post dose) (NL), n=58 | 34
  Day 2 (4 hours post dose) (Abn NCS), n=58 | 24
  Day 2 (4 hours post dose) (Abn CS), n=58 | 0
  Day 2 (8 hours post dose) (NL), n=58 | 30
  Day 2 (8 hours post dose) (Abn NCS), n=58 | 28
  Day 2 (8 hours post dose) (Abn CS), n=58 | 0
  Day 2 (12 hours post dose) (NL), n=58 | 31
  Day 2 (12 hours post dose) (Abn NCS), n=58 | 27
  Day 2 (12 hours post dose) (Abn CS), n=58 | 0
  Day 2 (24 hours post dose) (NL), n=58 | 34
  Day 2 (24 hours post dose) (Abn NCS), n=58 | 24
  Day 2 (24 hours post dose) (Abn CS), n=58 | 0
  Day 4 (Pre dose) (NL), n=56 | 31
  Day 4 (Pre dose) (Abn NCS), n=56 | 25
  Day 4 (Pre dose) (Abn CS), n=56 | 0
  Day 4 (4 hours post dose) (NL), n=55 | 26
  Day 4 (4 hours post dose) (Abn NCS), n=55 | 29
  Day 4 (4 hours post dose) (Abn CS), n=55 | 0
  Day 4 (8 hours post dose) (NL), n=55 | 25
  Day 4 (8 hours post dose) (Abn NCS), n=55 | 30
  Day 4 (8 hours post dose) (Abn CS), n=55 | 0
  Day 4 (12 hours post dose) (NL), n=55 | 27
  Day 4 (12 hours post dose) (Abn NCS), n=55 | 28
  Day 4 (12 hours post dose) (Abn CS), n=55 | 0
  Day 4 (24 hours post dose) (NL), n=54 | 28
  Day 4 (24 hours post dose) (Abn NCS), n=54 | 26
  Day 4 (24 hours post dose) (Abn CS), n=54 | 0
  Day 8-11 (NL), n=50 | 29
  Day 8-11 (Abn NCS), n=50 | 21
  Day 8-11 (Abn CS), n=50 | 0
  Follow-up (NL), n=2 | 1
  Follow-up (Abn NCS), n=2 | 1
  Follow-up (Abn CS), n=2 | 0

14. Secondary Outcome: Mean Area Under the Plasma Drug Concentration-time Curve (AUC) From Time Zero (Pre-dose) to the Last Time of Quantifiable Concentration (AUC[0-t]) and From Time Zero (Pre-dose) to 24 Hours Post Dose (AUC[0-24]) for Lapatinib
Description: AUC is defined as the area under the lapatinib concentration-time curve as a measure of drug exposure. AUC(0-t) and AUC(0-24) were determined from the plasma concentration-time data using the linear trapezoidal rule for increased concentrations and the logarithmic trapezoidal rule for decreased concentrations. For PK analysis, one blood sample was collected on Day 1 for placebo Baseline. The 24 hour blood sample on Day 2 also served for lapatinib Baseline. Pre-dose blood samples were collected 30 minutes prior to the administration of study medication on Day 2 (placebo) and Day 4 (lapatinib). Serial blood samples were collected on Day 2 (for placebo) and on Day 4 (for lapatinib) at the following post-last-dose time points 1, 2, 3, 4, 6, 8, 10, 12, and 24 hours.
Time Frame: Day 1 pre-dose; on Day 2 (at pre-dose, then 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post-last-dose), and on Day 4 (at pre-dose, then 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post-last-dose)
Population: Pharmacokinetic (PK) Population: all participants in the ATS Population for whom at least one PK sample was obtained and analyzed. Only participants available at the specified time point (represented as n=X in the category title) were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms hour per milliliter
Arm/Group | Lapatinib 2000 mg
Number analyzed (Participants) | 56
Nanograms hour per milliliter
  AUC[0-t]), n=56 | 56000 (73.4)
  AUC[0-24]), n=54 | 59200 (60.2)

15. Secondary Outcome: Mean Maximum Plasma Concentration (Cmax) and Observed Plasma Concentration at 24 Hours Post-dose (C24) of Lapatinib
Description: The first occurrence of Cmax and C24 was determined directly from the raw concentration-time data. For PK analysis, one blood sample was collected on Day 1 for placebo Baseline. The 24 hour blood sample on Day 2 also served for lapatinib Baseline. Pre-dose blood samples were collected 30 minutes prior to the administration of study medication on Day 2 (placebo) and Day 4 (lapatinib). Serial blood samples were collected on Day 2 (for placebo) and on Day 4 (for lapatinib) at the following post-last-dose time points 1, 2, 3, 4, 6, 8, 10, 12, and 24 hours.
Time Frame: Day1 pre-dose; on Day 2 (at pre-dose, then 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post-dose), and on Day 4 (at pre-dose, then 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post-dose)
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per mL
Arm/Group | Lapatinib 2000 mg
Number analyzed (Participants) | 56
Nanograms per mL
  Cmax, n=56 | 3920 (50.8)
  C24, n=54 | 1410 (88.1)

16. Secondary Outcome: Median Time to Cmax (Tmax) and the Time Prior to the First Quantifiable (Non-zero) Lapatinib Plasma Concentration (Tlag) Following the Last (3rd) Lapatinib Dose
Description: For each participant, the time at which Cmax was observed (tmax) was determined directly from the raw concentration-time data. For each participant, the time prior to the first quantifiable (non-zero) concentration (tlag) was determined directly from the raw concentration-time data. Since all participants received 2 doses of study medication prior to the collection of the first (pre-dose) blood sample on Day 4, tlag was expected to be zero. For PK analysis, one blood sample was collected on Day 1 for placebo Baseline. The 24 hour blood sample on Day 2 also served for lapatinib Baseline. Pre-dose blood samples were collected 30 minutes prior to the administration of study medication on Day 2 (placebo) and Day 4 (lapatinib). Serial blood samples were collected on Day 2 (for placebo) and on Day 4 (for lapatinib) at the following post-last-dose time points 1, 2, 3, 4, 6, 8, 10, 12, and 24 hours.
Time Frame: Day 1 pre-dose; on Day 2 (at pre-dose, then 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post-dose), and on Day 4 (at pre-dose, then 1, 2, 3, 4, 6, 8, 10, 12 and 24 hours post-dose)
Population: PK Population
Measure: Median (Full Range); unit: Hours
Arm/Group | Lapatinib 2000 mg
Number analyzed (Participants) | 56
Hours
  tmax | 3.55 [0 to 24.1]
  tlag | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from Day 1 until the follow-up visit (up to 28 days after the last dose of lapatinib [up to end of Study Week 4]).
Description: The number of participants in 1st Period - placebo (57) is different from 2nd Period - lapatinib (58) because one participant was "double dosed" with lapatinib (i.e., received lapatinib during both the 1st period and 2nd period) due to dosing error.
Arm/Group | Placebo | Lapatinib 2000 mg
Serious Adverse Events (participants affected / at risk) | 0/57 | 4/58
Other Adverse Events (participants affected / at risk) | 16/57 | 44/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=57) | Lapatinib 2000 mg (N=58)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=57) | Lapatinib 2000 mg (N=58)
Anaemia (Blood and lymphatic system disorders) | 0 | 9
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Conduction disorder (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 17
Dyspepsia (Gastrointestinal disorders) | 0 | 3
Nausea (Gastrointestinal disorders) | 4 | 5
Proctalgia (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 3
Chest pain (General disorders) | 1 | 1
Fatigue (General disorders) | 0 | 6
Mucosal inflammation (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 2
Cellulitis (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Rash pustular (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Dizziness (Nervous system disorders) | 1 | 2
Dysgeusia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Sinus headache (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 2
Hypotension (Vascular disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.